CLINICAL TRIAL: NCT02240758
Title: INTRA-OPERATIVE CONFOCAL LASER ENDOMICROSCOPY FOR BRAIN TUMORS: A FEASIBILITY STUDY IN HUMAN
Brief Title: Confocal Laser Endomicroscopy for Brain Tumors
Acronym: GLIOFOCAL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-820
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Low Grade Glioma (LGG), High Grade Glioma (HGG)
Keywords: glioma, confocal laser endomicroscopy
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgical removal of the tumors+stereotaxic biopsy (Experimental)
  Interventions: Procedure: confocal endomicroscopy with the CELLVIZIO® system (Mauna Kea technology)

INTERVENTIONS:
Procedure: confocal endomicroscopy with the CELLVIZIO® system (Mauna Kea technology) — The CELLVIZIO® system (Mauna Kea technology) will be used for confocal endomicroscopy during a surgical procedure (either open surgical approach or stereotaxic biopsy). The probe dedicated to the CELLVIZIO® system will be positioned against the surface of the brain, sequences will be acquired, and finally compared with anatomapathology exams. Two specific medications will be used as contrast agent in the study: Fluorescein FAURE 500mg/5mL IV with a maximum of two doses per patient OR 5 amino-levulinic hydrochloride (GLIOLAN, MEDAC) orally at the dose of 20mg/kg of body weight.

SUMMARY:
Confocal Laser Endomicroscopy (CLE) could be a useful tool for real-time diagnosis of brain lesions (initial diagnosis or follow-up post resection to check for residual dysplasia) and real-time assessment of resections margins during surgery. Probe-based CLE using the CELLVIZIO® has never been used for glioma surgical guided resection. Before assessing the potential of this technique in improving surgical resection outcome, a feasability study has to be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Clinical signs and history of the disease in favor of a HGG, LGG
* MRI study in favor of a HGG, LGG, meningioma or brain metastasis
* Affiliated to or beneficiary of a social security system (or equivalent).
* Patients who have provided written informed consent for the study

Exclusion Criteria:

* - Allergy to fluorescein
* Previous life-threatening allergic reactions and known hypersensitivity
* Pregnant or lactating or not using effective contraception;
* Restricted renal function define by a creatinine clearance < 30ml/min
* Patients under a beta-blockers treatment
* Contraindication to do an MRI (pace-maker)
* Contraindication to the use of 5-ALA : known hypersensibility to 5-ALA or to porphyrin, acute or chronic porphyria
* Minor or adult ward of court (under guardianship or trusteeship)
* No affiliation to a social security system (or equivalent).
* Patients who express opposition to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the technical feasibility of endomicroscopic imaging during brain tumors (gliomas) removal with an open approach (classic neurosurgical procedures) and biopsies. | End of the surgical procedure
  The technical feasibility will be assessed by the capacity of the CELLVIZIO® system to provide microscopic images of healthy tissue and lesions suspected with malignancy and to match those images with classical histologies.

SECONDARY OUTCOMES:
To demonstrate the safety of endomicroscopic imaging during brain tumors (gliomas, meningiomas, metastasis) removal with an open approach (classic neurosurgical procedures) and biopsies. | 14 days after inclusion
  Safety will be assessed by the number, type and severity of recorded adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: GUYOTAT JACQUES, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France